CLINICAL TRIAL: NCT04333537
Title: Randomized Phase II/III Trial of Sentinel Lymph Node Biopsy Versus Elective Neck Dissection for Early-Stage Oral Cavity Cancer
Brief Title: Comparing Sentinel Lymph Node (SLN) Biopsy With Standard Neck Dissection for Patients With Early-Stage Oral Cavity Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-HN006; NCI-2020-01542 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-HN006 (Other: NRG Oncology); NRG-HN006 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2020-03-26; First posted 2020-04-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Buccal Mucosa Squamous Cell Carcinoma; Floor of Mouth Squamous Cell Carcinoma; Gingival Squamous Cell Carcinoma; Hard Palate Squamous Cell Carcinoma; Lip Squamous Cell Carcinoma; Lower Alveolar Ridge Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma; Retromolar Trigone Squamous Cell Carcinoma; Stage I Lip and Oral Cavity Cancer AJCC v8; Stage II Lip and Oral Cavity Cancer AJCC v8; Tongue Squamous Cell Carcinoma; Upper Alveolar Ridge Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms | interventions — X-Rays; Fluorodeoxyglucose F18; acetyl-glycyl-asparagyl-glutaminyl-glutamyl-glutaminyl-valyl-seryl-prolyl-leucyl-threonyl-leucyl-leucyl-lysyl-lysyl-tryptophyl-cysteinyl-Alexa Fluoro 680 C2C2-maleimide conjugate; Neck Dissection; Magnetic Resonance Spectroscopy; Sentinel Lymph Node Biopsy; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (SLN biopsy) (Experimental): Patients receive an imaging agent via injection and undergo planar imaging and SPECT/CT over 1-2 hours. Patients then undergo SLN biopsy. Patients also undergo FDG PET/CT, CT, and/or chest x-ray at screening and during follow up.
  Interventions: Procedure: Chest Radiography; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Drug: Imaging Agent; Procedure: Planar Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Procedure: Sentinel Lymph Node Biopsy; Procedure: Single Photon Emission Computed Tomography
- Group II (END) (Active Comparator): Patients undergo standard END. Patients also undergo FDG PET/CT, CT, and/or chest x-ray at screening and during follow up.
  Interventions: Procedure: Chest Radiography; Other: Fludeoxyglucose F-18; Procedure: Neck Dissection; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Chest Radiography — Undergo chest x-ray
  Other Names: Chest X-ray
Procedure: Computed Tomography — Undergo SPECT/CT scan and FDG PET/CT or CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
  Arms: Group I (SLN biopsy)
Other: Fludeoxyglucose F-18 — Undergo FDG PET/CT
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Imaging Agent — Receive imaging agent via injection
  Other Names: Image Enhancement Agent
  Arms: Group I (SLN biopsy)
Procedure: Neck Dissection — Undergo standard elective neck dissection
  Arms: Group II (END)
Procedure: Planar Imaging — Undergo planar imaging
  Arms: Group I (SLN biopsy)
Procedure: Positron Emission Tomography — Undergo FDG PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Procedure: Sentinel Lymph Node Biopsy — Undergo SLN biopsy
  Other Names: Sentinel Node Biopsy; Sentinel node biopsy alone; SLNB; SNB
  Arms: Group I (SLN biopsy)
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT scan
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
  Arms: Group I (SLN biopsy)

SUMMARY:
This phase II/III trial studies how well sentinel lymph node biopsy works and compares sentinel lymph node biopsy surgery to standard neck dissection as part of the treatment for early-stage oral cavity cancer. Sentinel lymph node biopsy surgery is a procedure that removes a smaller number of lymph nodes from your neck because it uses an imaging agent to see which lymph nodes are most likely to have cancer. Standard neck dissection, such as elective neck dissection, removes many of the lymph nodes in your neck. Using sentinel lymph node biopsy surgery may work better in treating patients with early-stage oral cavity cancer compared to standard elective neck dissection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if patient-reported neck and shoulder function and related quality of life (QOL) at 6 months after surgery using the Neck Dissection Impairment Index (NDII) is superior with sentinel lymph node (SLN) biopsy compared to elective neck dissection (END) for treatment of early-stage oral cavity squamous cell carcinoma (OCSCC) (cT1-2N0). (Phase II) II. To determine if disease-free survival (DFS) is non-inferior with SLN biopsy compared to END for treatment of early-stage OCSCC (cT1-2N0). (Phase III) III. To determine if patient-reported neck and shoulder function and related QOL at 6 months after surgery using NDII is superior with SLN biopsy compared to END for treatment of early-stage OCSCC (cT1-2N0). (Phase III)

SECONDARY OBJECTIVES:

I. To compare patterns of failure (local-regional relapse and distant metastasis) between surgical arms.

II. To measure and compare overall survival (OS) between surgical arms. III. To measure and compare the toxicity of the two surgical arms.

IV. To measure longitudinal patient-reported neck and shoulder function and related QOL between surgical arms using the following instruments:

IVa. Neck Dissection Impairment Index (NDII); IVb. Abbreviated Disabilities of the Arm, Shoulder and Hand (QuickDASH); IVc. Functional Assessment of Cancer Therapy-Head and Neck (FACT-H&N). V. To assess the length of hospitalization, post-operative drain placement, and operative morbidity between arms.

VI. To estimate the negative predictive rate of fludeoxyglucose F-18 (FDG)-positron emission tomography (PET)/computed tomography (CT) for N0 neck in patients with T1 and T1-2 oral cavity squamous cell cancer (OCSCC) patients in the END arm.

VII. To assess nodal metastases rates between arms. VIII. To assess the pathologic false omission rate (FOR) in the SLN biopsy arm. IX. To determine if patient-reported neck and shoulder function using the NDII and related QOL at 6 months after surgery with SLN biopsy is superior to the END in low-risk patients.

X. To compare the diagnostic performance of planar only versus (vs.) single photon emission computed tomography (SPECT)/CT plus planar for SLN mapping (phase II only).

EXPLORATORY OBJECTIVES:

I. To compare changes in patient-reported outcomes (European Quality of Life Five Dimension Five Level Scale Questionnaire [EQ-5D-5L]) between surgical arms.

II. To collect biospecimens for future translational science studies. III. To assess the DFS between arms in low-risk patients.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive an imaging agent via injection and undergo planar imaging and SPECT/CT over 1-2 hours. Patients then undergo SLN biopsy. Patients also undergo FDG PET/CT, CT, and/or chest x-ray at screening and during follow up.

GROUP II: Patients undergo standard END. Patients also undergo FDG PET/CT, CT, and/or chest x-ray at screening and during follow up.

After completion of study treatment, patients are followed up 3 weeks after surgery, every 3 months for year 1, every 4 months for year 2, every 6 months for year 3, then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION INCLUSION:
* Pathologically (histologically or cytologically) proven diagnosis of squamous cell carcinoma (SCC) of the oral cavity, including the oral (mobile) tongue, floor of mouth (FOM), mucosal lip, buccal mucosa, lower alveolar ridge, upper alveolar ridge, retromolar gingiva (retromolar trigone; RMT), or hard palate prior to registration
* Appropriate stage for study entry (T1-2N0M0; American Joint Committee on Cancer [AJCC] 8th edition [ed.]) based on the following diagnostic workup:

  * History/physical examination within 42 days prior to registration
  * Imaging of head and neck within 42 days prior to registration

    * PET/CT scan or contrast neck CT scan, or gadolinium-enhanced neck magnetic resonance imaging (MRI) or lateral and central neck ultrasound; diagnostic quality CT is preferred and highly recommended as part of the PET/CT when possible
  * Imaging of chest within 42 days prior to registration

    * Chest x-ray, CT chest scan (with or without contrast), or PET/CT (with or without contrast)
* Surgical assessment within 42 days prior to registration. Patient must be a candidate for surgical intervention with sentinel lymph node (SLN) biopsy and potential completion neck dissection (CND) or elective neck dissection (END)

  * Surgical resection of the primary tumor will occur through a transoral approach with anticipation of resection free margins
* Age >= 18
* Zubrod performance status 0-2 within 42 days prior to registration
* For women of child-bearing potential, negative serum or urine pregnancy test within 42 days prior to registration
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
* Only patients who are able to read and understand English or French are eligible to participate as the mandatory patient reported NDII tool is only available in these languages
* PRIOR TO STEP 2 RANDOMIZATION:
* FDG PET/CT required prior to step 2. Note: FDG PET/CT done prior to step 1 can be submitted for central review

  * PET/CT node negative patients, determined by central read, will proceed to randomization. PET/CT node positive patients will go off study, but will be entered in a registry and data will be collected to record the pathological outcome of neck nodes for diagnostic imaging assessment and future clinical trial development

    * NOTE: All FDG PET/CT scans must be performed on an American College of Radiology (ACR) accredited scanner (or similar accrediting organization)
* The patient must complete NDII prior to step 2 registration

Exclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION EXCLUSION:
* Definitive clinical or radiologic evidence of regional (cervical) and/or distant metastatic disease
* Prior non-head and neck invasive malignancy (except non-melanomatous skin cancer, including effectively treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or cervix) unless disease free for ≥ 2 years
* Diagnosis of head and neck SCC in the oropharynx, nasopharynx, hypopharynx, and larynx
* Unable or unwilling to complete NDII (baseline only)
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for different cancer(s) is allowable
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Severe, active co-morbidity that would preclude an elective or completion neck dissection
* Pregnancy and breast-feeding mothers
* Incomplete resection of oral cavity lesion with a positive margin; however, an excisional biopsy is permitted
* Prior surgery involving the lateral neck, including neck dissection or gross injury to the neck that would preclude surgical dissection for this trial. Prior thyroid and central neck surgery is permissible; biopsy is permitted. Note: Borderline suspicious nodes that are >= 1 cm with radiographic finding suggestive of NOT malignant should be biopsied using ultrasound (U/S)-guided fine-needle aspiration (FNA) biopsy
* Underlying or documented history of hematologic malignancy (e.g., chronic lymphocytic leukemia [CLL]) or other active disease capable of causing lymphadenopathy (e.g., sarcoidosis or untreated mycobacterial infection)
* Actively receiving systemic cytotoxic chemotherapy, immunosuppressive, anti-monocyte or immunomodulatory therapy
* Currently participating in another investigational therapeutic trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2031-04-27 (Estimated); Study Completion 2031-04-27 (Estimated)

PRIMARY OUTCOMES:
Patient-reported neck and shoulder function (Phase II/III) | Before surgery (Baseline), 3 weeks after surgery, 3, 6, 12 months after surgery
  Will be evaluated and compared using the Neck Dissection Impairment Index (NDII), a 10-item tool between the two treatment arms. It is assumed that a 7.5-point between arm difference in the 6-month post-surgery NDII scores is clinically meaningful.
Patient reported quality of life (QOL) (Phase II) | Before surgery (Baseline), 3 weeks after surgery, 3, 6, 12 months after surgery
  Will be measured using 3 questionnaires over 12-15 minutes.
Disease-free survival (DFS) (phase III) | From randomization to local/regional recurrence, distant metastasis, or death due to any cause, whichever comes first, assessed up to 11 years
  Measured using Cox proportional hazards model and the Kaplan-Meier method. Failure includes local/regional recurrence, distant metastasis, or death due to any cause.

SECONDARY OUTCOMES:
Overall survival rate | From randomization to death due to any cause, assessed up to 11 years
  Will be estimated using the Kaplan-Meier method and between-arm differences compared using the log-rank test.
Loco-regional failure | From the time of randomization to the date of failure, date of precluding event, or last known follow-up date, assessed up to 11 years
  The cumulative incidence estimator will be used to estimate time to event distributions with between arm differences using cause-specific log-rank test.
Distant metastasis | From the time of randomization to the date of distant metastasis, date of precluding event, or last known follow-up date, assessed up to 11 years
  The cumulative incidence estimator will be used to estimate event distributions with between arm differences tested using cause-specific log-rank test.
Toxicity | Time of primary endpoint analysis
  Measured by the Common Terminology Criteria for Adverse Events version 5.0. The proportion of patients with at least 1 grade 3 or higher adverse event will be compared between treatment arms.
Patient-reported shoulder-related QOL, function impairment and disability | Baseline, 3 weeks, 3, 6, 12 months post-surgery
  Patient reported using Abbreviated Disabilities of the Arm, Shoulder, and Hand (QuickDASH) with scores of 0-100. A higher score indicates greater disability.
General quality of life | Baseline, 3 weeks, 3, 6, 12 months post-surgery
  Will be measured using the Functional Assessment of Cancer Therapy-Head and Neck to measure Functional Assessment of Cancer Therapy-Head and Neck-Trial Outcome Index scores on a scale from 0-96. A higher score indicates better quality of life.
Nodal metastasis detection rate | At time of surgery
  Defined as the proportion of patients with pathologic positive nodes using the pathology results.
Pathologic false omission rate | At time of surgery
  Measured within the sentinel lymph node biopsy (SLN) arm only. Defined as the proportion of patients with false negative results among negative SLN patients.
Length of hospital stay | Prior to surgery, at time of discharge from surgery
  Length of hospital stay due to surgical procedure will be compared between arms using the Mann-Whitney test.
Post-surgery patient-reported outcome | At 6 months post-surgery
  Measured by NDII in low-risk oral cavity squamous cell carcinoma patients using analysis of covariance comparison model.
Diagnostic performance (Phase II only) | Up to 11 years
  Descriptive statistics (minimum, maximum, mean, standard deviation, and coefficient of variation) of the number of detected SLNs will be calculated by modality and neck sublevel. The difference of the number of SLNs between single photon emission computed tomography/computed tomography plus planar and planar only will be computed and summarized by neck sublevel, reader, and overall. Pairwise absolute differences of the number of detected SLNs among readers will be computed and summarized by modality and neck sublevel.

OTHER OUTCOMES:
Quality of life | Baseline, 3 weeks, and 3, 6, 12 months post-surgery
  Measured by European Quality of Life Five Dimension Five Level Scale Questionnaire.
DFS for low-risk patients | From randomization to local/regional recurrence, distant metastasis, or death due to any cause, whichever comes first, assessed up to 11 years
  Exploratory analyses will be done using the Kaplan-Meier method to estimate the DFS distribution in both arms. Cox proportional hazards models with the treatment arm only and with treatment arms and relevant patient and tumor characteristics will be fitted. 95% confidence intervals (CIs) for the treatment effect from both models will be also reported.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Y Lai, Principal Investigator — NRG Oncology
Locations (100):
- United States (99):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Methodist Hospital, Memphis, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada